CLINICAL TRIAL: NCT00651690
Title: Study of Responsiveness of Seven Functional Tasks in Patients With Poststroke Upper Limb Spasticity With Botulinum Toxin Type A Treatment
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan, Inc.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 191622-065
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2008-05-28 (Estimated); Status verified 2008-05

CONDITIONS: Stroke; Muscle Spasticity
MeSH Terms: conditions — Stroke; Muscle Spasticity | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Botulinum Toxin Type A
  Interventions: Biological: Botulinum Toxin Type A
- 2 (Placebo Comparator): Saline
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Botulinum Toxin Type A — 200 U to 360 U of botulinum toxin Type A on Day 0. Patients who met retreatment criteria received a second treatment (open-label) at Week 12 or Week 18
  Other Names: BOTOX®
  Arms: 1
Biological: Placebo — Saline injection on Day 0
  Arms: 2

SUMMARY:
This study evaluates the responsiveness of 7 functional tasks to botulinum toxin Type A treatment in poststroke patients with spasticity of the upper-limb flexors

ELIGIBILITY:
Inclusion Criteria:

* Medically stable poststroke with focal unilateral upper-limb spasticity

Exclusion Criteria:

* Stroke within 6 months of the study enrollment visit
* Previous or current botulinum toxin therapy of any type in the study limb

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2004-03; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

PRIMARY OUTCOMES:
Seven functional tasks (nail filing, hand cleaning, holding a water bottle, brushing teeth, holding a small fruit, holding a medium fruit, and holding a large fruit) | Week 6

SECONDARY OUTCOMES:
Spasticity of the upper-limb flexors as measured by the Ashworth Scale | Week 6

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Indianapolis, Indiana, United States

REFERENCES:
- [Background] Turkel CC, Bowen B, Liu J, Brin MF. Pooled analysis of the safety of botulinum toxin type A in the treatment of poststroke spasticity. Arch Phys Med Rehabil. 2006 Jun;87(6):786-92. doi: 10.1016/j.apmr.2006.02.015. PMID 16731213
- [Background] Turkel C, Bowen B, Liu J, Brin M. A pooled analysis of the safety of BoNTA (BOTOX(R)) in the treatment of poststroke spasticity. Neurorehabil Neural Repair 2006;20(1):200 ABS-P3-081
- See also: Link to Clinical Trial Results — http://www.allerganclinicaltrials.com